CLINICAL TRIAL: NCT04076501
Title: Effect of Short-term Ambulatory Oxygen Therapy on Cardiopulmonary Exercise Capacity (CPET) in Patients With Grown-up Congenital Heart Disease (GUCH)
Brief Title: Effect of Short-term Oxygen During CPET in GUCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: KEK-ZH-NR. 2012-0251_4
Record Dates: First submitted 2019-08-30; First posted 2019-09-03 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Grown-up Congenital Heart Disease (GUCH)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplemental oxygen (Experimental): Supplemental oxygen will be applied via a mask during CPET
  Interventions: Procedure: Oxygen application
- Sham room air (Sham Comparator): Room air will be applied similarly to oxygen
  Interventions: Procedure: Sham room air

INTERVENTIONS:
Procedure: Oxygen application — Oxygen application Supplemental oxygen via mask
  Arms: Supplemental oxygen
Procedure: Sham room air — Room air applied via mask
  Arms: Sham room air

SUMMARY:
In a randomized, sham-controlled crossover trial the investigators will test whether supplemental oxygen given during cardiopulmonary exercise testing will improve exercise performance and physiological parameters in patients with grown-up congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* GUCH, stable medication for at least 4 weeks.

Exclusion Criteria:

* instable status, pregnancy, clinically relevant concomitant diseases, inability to follow the study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Work Rate (Watt) | 1 day
  Maximal Work Rate (Wmax) measured during cardiopulmonary exercise test oxygen vs. room air
Endurance Time (s) Endurance Time (s) Endurance Time (s) | 1 day
  Endurance (s) with 75% Wmax measured during cardiopulmonary exercise test oxygen vs. room air

SECONDARY OUTCOMES:
Peak Oxygen uptake | 1 day
  measured during cardiopulmonary exercise test oxygen vs. room air
Respiratory Exchange ratio | 1 day
  measured during cardiopulmonary exercise test oxygen vs. room air
Changes in arterial blood parameters | 1 day
  measured during cardiopulmonary exercise test oxygen vs. room air
muscle tissue oxygen | 1 day
  Oxygen saturation in the muscle measured during cardiopulmonary exercise test oxygen vs. room air with near infrared spectroscopy
cerebral tissue oxygen | 1 day
  Oxygen saturation in the brain measured during cardiopulmonary exercise test oxygen vs. room air with near infrared spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Division of Pneumology, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No